CLINICAL TRIAL: NCT03559582
Title: Diagnostics and Pharmacotherapy for Severe Forms of TB
Brief Title: Diagnostics and Pharmacotherapy for Severe Forms of TB (DMID 15-0100)
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Scientific Center for Family Health and Human Reproduction Problems, Russia (Other Government); Kilimanjaro Christian Medical Centre, Tanzania (Other); Haydom Lutheran Hospital (Other); Mbarara University of Science and Technology (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of Florida (Other)
Responsible Party: Principal Investigator, Scott Heysell, MD, Associate Professor of Medicine, Division of Infectious Diseases and International Health, University of Virginia
Other Study IDs: 18452; U01AI115594 (NIH)
Record Dates: First submitted 2018-02-22; First posted 2018-06-18 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will use clinical and related phenotypic data and saliva samples to identify and characterize genetic and molecular biological markers that will enrich our understanding of the biological basis of an individual's response to anti-TB drugs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major Research Aim: To study novel molecular diagnostics and the pharmacokinetic variability among a spectrum of TB disease states, including severe forms of TB like disseminated TB, TB meningitis and drug resistant TB, among adults and children from multiple international sites.

DETAILED DESCRIPTION:
Aim 1. Measure pharmacokinetics to anti-tuberculosis (TB) medications in severe TB syndromes (including multidrug-resistant TB, pediatric TB, TB sepsis and TB meningitis) from diverse geographies (including Tanzania, Uganda, Bangladesh, and Siberia) and correlate these findings to TB treatment outcome (TB treatment failure: death/ default/ relapse/ further acquired drug resistance).

Aim 2. Decipher mechanisms of pharmacokinetic variability to TB drugs, particularly malabsorption due to concurrent gastrointestinal disease.

Aim 3. Deployment of quantitative susceptibility testing (minimum inhibitory concentration-MIC) and rapid MIC-informed molecular methods (e.g., TaqMan Array Card-TAC) for M. tuberculosis.

In addition to the stated aims, the primary elements of capacity building requisite for this project include the training in and deployment of the fieldable molecular diagnostic platforms, onsite pharmacokinetic monitoring, and a broad strengthening of longitudinal cohort management for clinical research.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to one of the study site hospitals with at least ONE of the following:

1. Clinical suspicion for TB in a child, as defined by NIH Consensus Case Definitions for TB research in children, and started on TB treatment
2. Clinical suspicion for TB meningitis, as defined by the International TB Meningitis Workshop Consensus Case Definitions for TB Meningitis
3. Clinical suspicion for TB sepsis, as defined by the Uganda/PRISM-U definitions
4. Microbiologic evidence of MDR-TB from a respiratory specimen within the past 6 months

Exclusion Criteria:

1. Pregnant women-self reported
2. Patient unable per treating physician discretion to undergo sample collection
3. Patient or representative/guardian unable to sign written informed consent
4. Patient unable to return for follow-up or be contacted by phone for follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited by medical officer review of new admissions to the TB hospitals at the study sites- Kibong'oto National TB Hospital (Tanzania), Haydom Lutheran Hospital (Tanzania), Irkutsk Regional Clinical Tuberculosis Hospital (Siberia/Russian Federation), National Institute of Diseases of the Chest Hospital (Bangladesh), ICDDRB Hospital (Bangladesh), Mbarara Regional Referral Hospital (Uganda).
Sampling Method: Non-Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Measure area under the concentration curve (AUC) to anti-tuberculosis (TB) medications relative to TB treatment outcome in severe TB syndromes | December 2019
  Severe TB syndromes include multidrug-resistant TB, pediatric TB, TB sepsis and TB meningitis from diverse geographies (including Tanzania, Uganda, Bangladesh, and Siberia). The parameter of most importance to cidal activity of anti-TB medications among the cohort is AUC. TB treatment outcome will be defined as death, microbiological failure, relapse or acquired drug resistance, and machine learning algorithms such as classification and regression tree analyses will be used to define AUC threshold for each anti-TB medication predictive of poor TB treatment outcome. Conventional logistic regression will then be used to determine the additive odds for a patient with one of more medications below an algorithm derived threshold being significantly more likely to have a poor TB treatment outcome.

SECONDARY OUTCOMES:
Collect stool in patients undergoing pharmacokinetic testing to measure the environmental enteropathy index | December 2019
  Stool will be collected in patients with severe TB syndromes undergoing pharmacokinetic testing and assayed for stool biomarkers of malabsorption (environmental enteropathy index) and modeled as a determinant of those with AUC values of one or more anti-TB medications below thresholds predictive of TB treatment outcome.
Collect stool in patients undergoing pharmacokinetic testing to measure the quantitative burden and species distribution of enteric pathogens by the enteric TAC assay- 35 bacterial, viral, parasitic species) | December 2019
  Stool will be collected in patients with severe TB syndromes undergoing pharmacokinetic testing and assayed for detection of molecular targets of enteric pathogens by TaqMan Array Card (TAC) platform. Enteric pathogen burden (including the effect of multiple pathogens in a single sample) will be modeled as a determinant of those with AUC values of one or more anti-TB medications below thresholds predictive of TB treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Heysell, MD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heysell SK, Mpagama SG, Ogarkov OB, Conaway M, Ahmed S, Zhdanova S, Pholwat S, Alshaer MH, Chongolo AM, Mujaga B, Sariko M, Saba S, Rahman SMM, Uddin MKM, Suzdalnitsky A, Moiseeva E, Zorkaltseva E, Koshcheyev M, Vitko S, Mmbaga BT, Kibiki GS, Pasipanodya JG, Peloquin CA, Banu S, Houpt ER. Pharmacokinetic-Pharmacodynamic Determinants of Clinical Outcomes for Rifampin-Resistant Tuberculosis: A Multisite Prospective Cohort Study. Clin Infect Dis. 2023 Feb 8;76(3):497-505. doi: 10.1093/cid/ciac511. PMID 35731948